CLINICAL TRIAL: NCT07292493
Title: The Role of Complement in Diabetic Kidney Disease
Brief Title: Immune System in Diabetic Kidney Disease
Acronym: KID-CODE
Status: Enrolling by invitation | Type: Observational
Sponsor: University Medical Centre Ljubljana (Other)
Responsible Party: Sponsor
Other Study IDs: 20250187
Record Dates: First submitted 2025-11-19; First posted 2025-12-18 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-11

CONDITIONS: Diabetes; Diabetic Kidney Disease; Complement System
Keywords: diabetes; diabetic kidney disease; complement system; C3; CD59; MAC; MBL; C3a; C3b; C5a; new antidiabetic drugs
MeSH Terms: conditions — Diabetes Mellitus; Diabetic Nephropathies; Complement Component 3 Deficiency, Autosomal Recessive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Patients with type 1 diabetes without chronic kidney disease: The investigators will include male and female patients aged between 40 and 65 years, who have diagnosis of diabetes for at least 10 years and no more than 25 years, with a body mass index below 30 kg/m², and without known macrovascular complications (coronary artery, peripheral arterial, or cerebrovascular disease). All participants must be treated with angiotensin-converting enzyme inhibitors or angiotensin receptor blockers at the highest tolerated dose. Individuals without known chronic kidney disease must meet kidney function criteria with an estimated glomerular filtration rate (eGFR) ≥ 60 ml/min and a urine albumin-to-creatinine ratio (UACR) < 3 g/mol.
- Patients with type 1 diabetes and chronic kidney disease: The investigators will include male and female patients aged between 40 and 65 years, who have diagnosis of diabetes for at least 10 years and no more than 25 years, with a body mass index below 30 kg/m², and without known macrovascular complications (coronary artery, peripheral arterial, or cerebrovascular disease). All participants must be treated with angiotensin-converting enzyme inhibitors or angiotensin receptor blockers at the highest tolerated dose. Individuals diagnosed with chronic kidney disease must meet the criteria of kidney function eGFR < 60 ml/min and UACR > 3 g/mol, or UACR > 30 g/mol regardless of eGFR.
- Patients with type 2 diabetes and chronic kidney disease: The investigators will include male and female patients aged between 40 and 65 years, who have diagnosis of diabetes for at least 10 years and no more than 25 years, with a body mass index below 30 kg/m², and without known macrovascular complications (coronary artery, peripheral arterial, or cerebrovascular disease). All participants must be treated with angiotensin-converting enzyme inhibitors or angiotensin receptor blockers at the highest tolerated dose. Individuals diagnosed with chronic kidney disease must meet the criteria of kidney function eGFR < 60 ml/min and UACR > 3 g/mol, or UACR > 30 g/mol regardless of eGFR.

SUMMARY:
Diabetes is a chronic condition marked by long-term elevated blood glucose levels. There are more types of diabetes; the majority of patients have type 1 or type 2 diabetes. Over long period of time, high blood sugar damages blood vessels and organs. One of the most common complications is diabetic kidney disease, which can slowly lead to kidney failure. People with this condition also have a much higher risk of heart and blood vessel diseases.

Newer research shows that the immune system, especially the complement system (a group of proteins that help defend the body), may also play a role in worsening kidney disease in diabetes. High blood sugar can activate these proteins, and they have been found in kidney tissue of patients with diabetic kidney disease.

The goal of this study is to find out how much the complement system contributes to kidney damage in diabetes, whether it affects different groups of patients differently, and whether it is linked to blood vessel health or the stage of kidney disease. The study will also assess if improved diabetes control is linked to reduced complement system activity.

DETAILED DESCRIPTION:
Diabetes is a chronic disease characterized by long-term elevated blood glucose levels. Several types of diabetes are known, with most affected individuals having type 1 or type 2 diabetes. Long-term elevation of blood glucose affects various organs in the body, a condition referred to as chronic complications of diabetes. Since elevated blood glucose damages both small and large blood vessels, complications are classified as microvascular (damage to small vessels) and macrovascular (damage to large vessels). Diabetic kidney disease is the main microvascular complication in both type 1 and type 2 diabetes and is also the leading cause of kidney failure.

Changes in the kidneys develop over many years. Gradual deterioration of kidney function is monitored using laboratory parameters. Along with declining kidney function, blood pressure also increases, and cardiovascular diseases begin to develop- the risk of these rises exponentially with worsening kidney function. Cardiovascular diseases represent the leading cause of mortality among people with diabetes.

Traditionally, diabetic kidney disease was considered as non-inflammatory condition. Its development was attributed to impaired glucose metabolism and elevated blood pressure. Consequently, achieving optimal blood glucose and blood pressure values has been regarded as key to preventing chronic complications. However, diabetes itself represents an additional risk factor for cardiovascular disease compared with individuals without diabetes. Thus, individuals with diabetic kidney disease are even more prone to cardiovascular events. In these patients it is especially important to follow treatment guidelines and to treat elevated blood glucose and blood pressure as intensively as possible. For individuals with diabetic kidney disease, medications from the group of angiotensin-converting enzyme inhibitors or angiotensin receptor blockers are prescribed for the treatment of high blood pressure. Both medication groups also have a protective effect on the kidneys and slow the decline of kidney function. Angiotensin is a substance in the body responsible for raising blood pressure-when its action is inhibited, blood pressure decreases.

The investigators now know that inflammation and the immune system also play a role in the development of chronic diabetic complications. The complement system (a group of proteins in the blood involved in immune responses) is becoming recognized for its importance. Current studies do not suggest that the complement system plays a key role in the onset of the disease; however, its role in the progression of diabetic kidney disease and possibly in the occurrence of different forms of the disease has become evident. Hyperglycaemia increases the activity of certain complement proteins and activates specific pathways, while the hyperglycaemic environment also impairs the regulation of some proteins. Kidney biopsies of individuals with diabetic kidney disease have shown the presence of complement proteins in kidney tissue, and gene expression analyses have identified activation of complement-related genes.

The purpose of this study is to determine whether and to what extent activation of the complement system contributes to diabetic kidney disease and to define potential differences among different groups of individuals with diabetes. Additionally, the investigators aim to determine whether there is a connection between complement system activation and arterial function, as well as between complement system activation and the stage of kidney disease. The investigators will also investigate whether diabetes control influences complement system activation and whether previous kidney biopsy findings correspond with laboratory results.

ELIGIBILITY:
Inclusion Criteria:

* body mass index below 30 kg/m²
* unknown macrovascular complications
* treated with angiotensin-converting enzyme inhibitors or angiotensin receptor blockers at the highest tolerated dose

Exclusion Criteria:

* a body mass index above 30 kg/m²
* macrovascular complications

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with type 1 and type 2 diabetes, who are being treated at the diabetology outpatient clinic of the Department of Endocrinology, Diabetes, and Metabolic Diseases, University Medical Centre Ljubljana.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Level of complement system activation | An additional visit to the diabetes outpatient clinic is planned within one year, where this will be determined.
  The investigators will determine components of the complement system in blood and urine samples.
  * Blood parameters:
    * complement component C3 - (expressed in g/L),
    * complement component C4 - (expressed in g/L),
    * factor B - (expressed in mg/L)
    * factor H - (expressed in mg/L),
    * factor I - (expressed in mg/L),
    * SC5b-9 lytic complex - (expressed in µg/L),
    * factor B fragment(Bb) - (expressed in µg/L),
    * factor H antibodies - (expressed in U/mL),
    * C1q Antibodies - (expressed in U/mL),
    * complement component C3a - (expressed in µg/L),
    * complement component C3c - (expressed in mg/L),
    * complement component C5a - (expressed in µg/L).
  * Urine parameter :
    * SC5b-9 lytic complex (expressed in µg/L)

SECONDARY OUTCOMES:
IMT thickness | An additional visit to the diabetes outpatient clinic is planned within one year, where the examination will be performed.
  The investigators will measure the intima-media thickness (IMT) with ultrasound. Result will be expressed in millimetres.
Carotid-femoral pulse wave velocity (PWV) | An additional visit to the diabetes outpatient clinic is planned within one year, where the examination will be performed.
  The investigators will evaluate arterial stiffness and central hemodynamics non-invasively using applanation tonometry and pulse wave analysis. Results will be expressed in metres per second (m/s).
Endothelial Function | An additional visit to the diabetes outpatient clinic is planned within one year, where the examination will be performed.
  The investigators will use peripheral arterial tonometry . The measurement is performed using a finger-mounted pneumatic probe, which detects pulsatile volume changes in the fingertip. The device's software analyses the change in pulse amplitude before and after occlusion, calculating the Reactive Hyperemia Index (RHI), which serves as a quantitative marker of endothelial function and has no unit.

CONTACTS AND LOCATIONS:
Overall Officials: Miodrag Janić, Principal Investigator
Locations (1):
- University Medical Centre Ljubljana, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Li MR, Sun ZJ, Chang DY, Yu XJ, Wang SX, Chen M, Zhao MH. C3c deposition predicts worse renal outcomes in patients with biopsy-proven diabetic kidney disease in type 2 diabetes mellitus. J Diabetes. 2022 Apr;14(4):291-297. doi: 10.1111/1753-0407.13264. Epub 2022 Mar 24. PMID 35322566
- [Background] Ostergaard JA, Thiel S, Lajer M, Steffensen R, Parving HH, Flyvbjerg A, Rossing P, Tarnow L, Hansen TK. Increased all-cause mortality in patients with type 1 diabetes and high-expression mannan-binding lectin genotypes: a 12-year follow-up study. Diabetes Care. 2015 Oct;38(10):1898-903. doi: 10.2337/dc15-0851. Epub 2015 Jul 15. PMID 26180106
- [Background] Hansen TK, Tarnow L, Thiel S, Steffensen R, Stehouwer CD, Schalkwijk CG, Parving HH, Flyvbjerg A. Association between mannose-binding lectin and vascular complications in type 1 diabetes. Diabetes. 2004 Jun;53(6):1570-6. doi: 10.2337/diabetes.53.6.1570. PMID 15161763
- [Background] Flyvbjerg A. The role of the complement system in diabetic nephropathy. Nat Rev Nephrol. 2017 May;13(5):311-318. doi: 10.1038/nrneph.2017.31. Epub 2017 Mar 6. PMID 28262777